CLINICAL TRIAL: NCT01161589
Title: First Arrhythmia Collection of Transvenous and Simultaneous Subcutaneous Implantable Defibrillator Data
Acronym: FACTS
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Linda Smith, Cameron Health
Other Study IDs: FACTS S-ICD
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Atrial Fibrillation
Keywords: sensing; S-ICD; ICD; CRT D
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical study is to collect simultaneous, multiple view cardiac signals representing both transvenous ICDs (T-ICD) and sensing vectors from the subcutaneous implantable defibrillator system (S-ICD). Upon completion, this data will represent the first true database capable of comparing detection characteristics of transvenous and subcutaneous ICDs. Future protocols will be created to dictate the specific methods of such comparisons.

DETAILED DESCRIPTION:
The FACTS S-ICD study is a data gathering study that takes place during the implant procedure of a standard T-ICD system. Patients undergoing a routine dual chamber, dual high voltage shocking coil T-ICD or CRT-D insertion or replacement will be connected to an external data recorder via sterile cables. Atrial and ventricular arrhythmias will be induced while multiple ECG views are simultaneously recorded from both intracardiac and surface vectors. These episodes will then be digitized to create the FACTS S-ICD arrhythmia library.

As both dedicated and integrated bipolar sensing configurations are currently utilized in the marketplace, data will be collected using both market available ICD sensing methods.

The FACTS S-ICD study will enroll a sufficient quantity of patients such that a minimum of 50 atrial and 50 ventricular arrhythmic episodes are collected via both dedicated and integrated ICD systems. S-ICD signals will be collected for all recorded episodes.

The T-ICD implant procedure will be completed as per normal hospital practice and no further patient dependent data gathering will be required past the implant surgery and point of surgery arrhythmia inductions.

INCLUSION CRITERIA

1. Age 18 or above, or legal age to give consent specific to state and national law.
2. Any patient undergoing a clinically indicated initial dual chamber T-ICD or CRT-D implantation. In addition, patients who require replacement of an existing dual chamber T-ICD or CRT-D system will be eligible for enrollment in the study.
3. Patient will have a subcutaneous, left pectoral defibrillator implant.

EXCLUSION CRITERIA

1. Patients unable or unwilling to provide informed consent.
2. Any condition which precludes the subject's ability to comply with the study requirements, including completion of the study.
3. Patients in chronic atrial fibrillation who have not been in sinus rhythm within the last six months.
4. Enrollment in a concurrent study, without Cameron Health's written approval, that may confound the results of this study.
5. Women who are pregnant or who are trying to become pregnant Note: Women of child bearing potential must have a negative pregnancy test within 7 days prior to defibrillator implant.
6. Patient requires left sub-muscular or right sided defibrillator implant

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or legal age to give consent specific to state and national law.
* Any patient undergoing a clinically indicated initial dual chamber T-ICD or CRT-D implantation. In addition, patients who require replacement of an existing dual chamber T-ICD or CRT-D system will be eligible for enrollment in the study.
* Patient will have a subcutaneous, left pectoral defibrillator implant

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent.
* Any condition which precludes the subject's ability to comply with the study requirements, including completion of the study.
* Patients in chronic atrial fibrillation who have not been in sinus rhythm within the last six months.
* Enrollment in a concurrent study, without Cameron Health's written approval, that may confound the results of this study.
* Women who are pregnant or who are trying to become pregnant Note: Women of child bearing potential must have a negative pregnancy test within 7 days prior to defibrillator implant.
* Patient requires left sub-muscular or right sided defibrillator implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a routine dual chamber, dual high voltage shocking coil T-ICD or CRT-D insertion or replacement
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Collection of simultaneous cardiac signals representing S-ICD and ICD sensing vectors | 3 years
  This study will enroll a sufficient number of patients such that a minimum of 50 atrial and 50 ventricular arrhythmic episodes are collected by dedicated and integrated ICD systems and by the simulated S-ICD system

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- Erasmus Medical Centre, Rotterdam, Netherlands